CLINICAL TRIAL: NCT03196024
Title: A Randomized Controlled Trial to Examine a Healthy Lifestyle Intervention With Families to Prevent Cardiovascular Disease and Type 2 Diabetes in Hispanics/Latinos
Brief Title: Corazon de la Familia (Heart of the Family)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Mudd (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Gia Mudd, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01NR016262-01A1 (NIH); 1R01NR016262-01A1 (NIH)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Risk Reduction Behavior; Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Diabetes; CVD; Lifestyle; Hispanic; Promotora; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Risk Reduction Behavior; Hispanic Americans; Latinos; Community Health Workers
MeSH Terms: conditions — Risk Reduction Behavior; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized controlled trial with Hispanic family dyads using a 2-group design (Corazón de la Familia active intervention versus control condition) to test effects of a type 2 diabetes and CVD risk reduction intervention at 3 (short-term) and 12 (long-term) months. For dyads randomized to the active intervention, the participant with 2 or more CVD or type 2 diabetes risk factors (index participant) and their co-participating family member will attend 8 sessions that provide type 2 diabetes and CVD risk reduction and lifestyle modification education. For dyads randomized to the control condition, only the index participant will attend 8 educational lifestyle modification sessions. Participants in both groups will receive monthly follow up phone calls up through 12 months post-baseline. The sessions for both the intervention and the control group and the monthly post-intervention phone calls will be provided by community health workers.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, community health workers, and assessors are blinded to which arm is the active intervention and which arm is the active comparator. Participants, community health workers, and assessors will be blinded to hypotheses regarding group differences and will be informed that both groups are intervention groups and that we are examining how well both intervention types perform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-focused intervention arm (Experimental): Family-focused intervention arm: Educational sessions will be provided to family pairs that include participants who are at-risk for type 2 diabetes or CVD and their co-participating family member.
  Interventions: Behavioral: Family-focused intervention arm
- Individual-focused intervention arm (Active Comparator): Individual-focused intervention arm: Educational sessions will be provided to the individual members of the family pairs who are at-risk for type 2 diabetes or CVD.
  Interventions: Behavioral: Individual-focused intervention arm

INTERVENTIONS:
Behavioral: Family-focused intervention arm — Family pairs including an individual family member at-risk for type 2 diabetes or CVD and a co-participating family member will be enrolled in the study. After completing baseline data they will be randomly selected to participate in one of the two study arms. For the family-focused arm, the family pair will attend 8 2-hour weekly educational sessions about type 2 diabetes and CVD risk reducing lifestyle behaviors. The sessions will be presented by community health workers (CHWs) in Spanish to groups of 5 to 6 family pairs. Following completion of the sessions, data will be collected from the family pairs. CHWs will call monthly to provide information and support through the end of the 12-month period at which time data will be collected from the family pairs.
  Arms: Family-focused intervention arm
Behavioral: Individual-focused intervention arm — Family pairs including an individual family member at-risk for type 2 diabetes or CVD and co-participating family member will be enrolled in the study. After completing baseline data pairs will be randomly selected to participate in one of two interventions. For the individual-focused intervention, the at-risk individual will attend 8 weekly 2-hour education sessions on type 2 diabetes and CVD risk reducing lifestyle behaviors. Sessions will be presented by CHWs in Spanish to groups of 10 to 12 individuals. Following completion of sessions, data will be collected from the individuals. CHWs will call monthly to provide information and support through the end of the 12-month period at which time data will be collected from the at-risk individuals and their co-participating family members.
  Arms: Individual-focused intervention arm

SUMMARY:
The Corazón de la Familia study is a randomized controlled trial to examine the effects of a novel family-focused lifestyle modification intervention to reduce risk for type 2 diabetes and cardiovascular disease (CVD) among Hispanics/Latinos. Facilitated by community health workers, the family-focused intervention engages two members of a family in an educational program addressing lifestyle behaviors to support sustained engagement in healthy lifestyles among Hispanics with high risk for type 2 diabetes or CVD. In this study, we will conduct a randomized controlled trial using a 2-group design and compare the short-term and long-term impact of the family-focused active intervention to an individual-focused control condition on biological and behavioral type 2 diabetes and CVD risk factors. Furthermore, we will examine outcomes of participants in the family-focused intervention to determine how each family member's engagement in healthy lifestyle behaviors and level of support for the other family member's engagement in healthy lifestyle behaviors affects their own and their partner's outcomes.

DETAILED DESCRIPTION:
The Corazón de la Familia study is a randomized controlled trial conducted to examine if a novel family-focused lifestyle modification intervention is more effective in reducing risk for type 2 diabetes and cardiovascular disease (CVD) than an individual-focused lifestyle modification intervention. We will enroll 220 Hispanic family pairs or dyads, of whom one member has two or more risk factors for type 2 diabetes or CVD but does not have type 2 diabetes or CVD. The second member of the family dyad may or may not have type 2 diabetes or CVD or may or may not be at risk for type 2 diabetes or CVD. Of the 220 family dyads, 110 will be randomly selected to participate in the family-focused intervention and 110 will be randomly selected to participate in the individual-focused intervention. The interventions for both groups will be provided by community health workers. Both groups will receive eight educational sessions about healthy lifestyle behaviors and support to address personal and environmental barriers to engaging in healthy behaviors. After the eight sessions, the community health workers will follow up with participants once a month by phone over the next 12 months. Primary outcomes include short-term and long-term impact of the family-focused active intervention compared to the individual-focused control condition on type 2 diabetes and CVD biological risk factors (for example, blood pressure and weight) and behavioral risk factors (for example, physical activity and tobacco use). Outcomes are measured at baseline, immediately post-intervention, and at the end of the 12 month period of the study for both groups.

ELIGIBILITY:
Inclusion Criteria:

We are enrolling family dyads, or 2 family members, one of whom is at-risk for type 2 diabetes or cardiovascular disease and the second of whom is a co-participating family member who may or may not be at risk for type 2 diabetes or cardiovascular disease.

Inclusion criteria for the at-risk member of the dyad:

* Is Hispanic or Latino
* Is 18 years of age and older
* Is a primary Spanish speaker
* Has two or more risk factors for type 2 diabetes or cardiovascular disease including:

  1. clinical diagnosis of hypertension;
  2. clinical diagnosis of hyperlipidemia;
  3. clinical diagnosis of prediabetes;
  4. overweight or obese (body mass index ≥ 25 kg/m2);
  5. is a current cigarette smoker;
  6. male 45 years of age or older or female 55 years of age or older;
  7. family history in first degree relative of type 2 diabetes or cardiovascular disease; or
  8. is a female with a history of gestational diabetes mellitus or polycystic ovary syndrome.
* Plan to be in Kentucky and Is willing to participate in the study for the next 12 months

Inclusion criteria for the co-participating member of the dyad

* Is 18 years of age and older
* At a minimum, understands Spanish
* Lives in the same household or in close proximity (no further than 25 miles distance) to the at-risk member of the dyad

Exclusion Criteria:

Exclusion criteria for family dyads:

* Dyads will be excluded if one or both dyad members have any of the following:
* Have cognitive impairment that preclude them from understanding the consent process, answering questionnaires, or participating in the intervention;
* Have a major psychiatric (e.g., schizophrenia) condition;
* Are pregnant or nursing or plan on becoming pregnant within the next year since dietary needs will be different.

Exclusion criteria that apply only to the at-risk member of the dyad:

* Have known coronary artery or cerebrovascular disease;
* Have a diagnosis of type 1 or type 2 diabetes;
* Have medical contraindications to participate in a lifestyle intervention that includes unsupervised physical activity and weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | Baseline, 3 months, and 12 months
  BMI based on measurements of weight and height and calculated as kg/m2
Change in blood pressure | Baseline, 3 months, and 12 months
  Blood pressure assessed using calibrated sphygmomanometry
Change in lipid profile | Baseline, 3 months, and 12 months
  Lipid profile includes LDL-cholesterol, HDL-cholesterol and triglycerides measured using point-of-care testing obtained by fingerstick.
Change in hemoglobin A1c (HbA1c) | Baseline, 3 months, and 12 months
  HbA1c measured using point-of-care testing obtained by fingerstick.
Change in level of physical activity | Baseline, 3 months, and 12 months
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ) to assess the number of days in the last 7 days that the participant engaged in vigorous or moderate physical activity and confirmed by comparing responses to number of daily steps over 7 days assessed with a Fitbit
Change in diet quality | Baseline, 3 months, and 12 months
  Diet quality will be measured using the Food Frequency Questionnaire
Change in tobacco use | Baseline, 3 months, and 12 months
  Urine cotinine levels will be used to assess tobacco use

SECONDARY OUTCOMES:
Support for healthy behaviors | Baseline, 3 months, and 12 months
  Self report of experience of social support for healthy behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gia Mudd-Martin, PhD, RN, Principal Investigator — University of Kentucky; Rosa Martin, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study will be made available after completion of analyses for primary and secondary outcomes, and publications and research presentations that address the specific aims and major secondary analyses of the study. Data will be submitted to the Inter-university Consortium for Political and Social Research (ICPSR), a unit of the Institute for Social Research at the University of Michigan. The PI will remove all direct and indirect identifiers from the study data before submitting data to ICPSR. The ICPSR also carefully reviews submitted datasets to assure confidentiality of human subjects is preserved. All de-identified data housed by ICPSR are available to over 759 member institutions as well as to other institutions and individuals. Should access to data from this study be restricted to member institutions, the PI will, on request, provide the de-identified dataset and accompanying documentation to requesters.
Time Frame: De-identified data from this study will be made available after completion of analyses for primary and secondary outcomes, and publications and research presentations that address the specific aims and major secondary analyses of the study.
Access Criteria: De-identified data from this study will be submitted to the Inter-university Consortium for Political and Social Research (ICPSR), a unit of the Institute for Social Research at the University of Michigan.All de-identified data housed by ICPSR are available to over 759 member institutions as well as to other institutions and individuals. Should access to data from this study be restricted to member institutions, the PI will, on request, provide the de-identified dataset and accompanying documentation to requesters.

DOCUMENTS (1):
  • Informed Consent Form (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03196024/ICF_000.pdf